CLINICAL TRIAL: NCT02368574
Title: Comparison of Class II and Class III Hysterectomy in Early Stage Cervical Cancer Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Gynecological Oncology Group (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGOG-001
Record Dates: First submitted 2015-01-18; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Class III hysterectomy Arm (No Intervention): Class III hysterectomy (radical hysterectomy): This procedure may be performed through laparotomy or laparoscope. Perivesical space and perirectal space should be opened, and the ureteral tunnel is completely separated and pushed down to the junction of ureter and urinary bladder. The uterine arteries are ligated at the level of internal iliac artery, and all the supporting ligaments and connective tissues around the uterus should be separated and abscised. The uterosacral ligament is removed near the sacrum, the cardinal ligament is removed near the pelvic wall, and the vagina is removed after the excision of peivaginal connective tissues, about 3-4cm from the cervical lesion. The pelvic lymph nodes are usually dissected at the same time.
- Class II hysterectomy Arm (Experimental): Class II hysterectomy (modified radical hysterectomy): This procedure may be performed through laparotomy or laparoscope. The scope of surgery is more extensive than Class I epifascial panhysterectomy, demanding the excision of more parametrium but reservation of the blood supply for distal ureter and urinary bladder. The ureter is separated from the ureteral tunnel, the vesicouterine ligament should be intact, and 1/2 uterosacral ligament and 1cm vagina are excised. The pelvic lymph nodes are usually dissected at the same time.
  Interventions: Procedure: Class II hysterectomy

INTERVENTIONS:
Procedure: Class II hysterectomy — Class II hysterectomy
  Arms: Class II hysterectomy Arm

SUMMARY:
Based on the value-based medicine, a randomized clinical trial was conducted to compare the role of class II and class III hysterectomy in patients with low risk early staged cervical cancer (defined as tumor lesions less than 2cm with less than 50% stromal invasion).

DETAILED DESCRIPTION:
This is a 1:1 multi-center randomized trial with class II hysterectomy plus node dissection as the experimental arm, and class III hysterectomy plus pelvic node dissection as the control arm. Primary endpoints are: (1). 3-year diseases-free survival (DFS) rate; (2) the rates of treatment-related toxicity; (3) post-operation QoL (including sexual function) and (4) treatment costs. Secondary endpoints are：(1) the rates of pelvic and/or extra-pelvic relapse; (2) overall survival(OS) rate; (3) the numbers of retroperitoneal node dissection, and (4) the rates of parametrial, margins and pelvic/para-aortic nodes involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IA2 and small IB1 <2 cm
2. Less than 50% stromal invasion based on MRI OR 10mm stromal invasion based on the pathology measurement of the LEEP/cone specimen
3. Squamous OR adenocarcinoma OR adenosquamous
4. Grade 1, 2 and 3
5. Lymph-vascular space invasion (LVSI): presence or absence
6. Diagnosis confirmed by LEEP/cone/cervical biopsy
7. Pelvic MRI in patients with involved cone/LEEP margins and those who had cervical biopsy only
8. Abdomino-pelvic CT scan in patients with negative LEEP-cone margins
9. No contraindications to surgery
10. No desire to preserve fertility
11. Informed consent

Exclusion Criteria:

1. High-risk histology types (clear cell, small cell etc)
2. Evidence of lymph node metastasis on preoperative imaging
3. Stage 1A1
4. Neo-adjuvant chemotherapy
5. Pregnancy
6. Desire to preserve fertility

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival (DFS) rate | up to 4 years

SECONDARY OUTCOMES:
Treatment-related toxicity | up to 4 years
Post-operation quality of life | up to 4 years
Cost effective | up to 4 years
Pelvic and/or extra-pelvic relapse rate | up to 4 years
Overall survival | up to 4 years
Node number involved in retroperitoneal node dissection | up to 4 years
Rates of parametrial, margins and pelvic/para-aortic nodes involvement | up to 4 years

REFERENCES:
- [Derived] Sun H, Cao D, Shen K, Yang J, Xiang Y, Feng F, Wu L, Zhang Z, Ling B, Song L. Piver Type II vs. Type III Hysterectomy in the Treatment of Early-Stage Cervical Cancer: Midterm Follow-up Results of a Randomized Controlled Trial. Front Oncol. 2018 Nov 28;8:568. doi: 10.3389/fonc.2018.00568. eCollection 2018. PMID 30555800